CLINICAL TRIAL: NCT03970915
Title: Evaluation of Warm-up Efficiency by Body Warmer Versus Standard Procedure in Severely Traumatized Patients During Pre-hospital Medical Management
Brief Title: Warm-up Efficiency by Body Warmer Versus Standard Procedure in Severely Traumatized Patients
Acronym: THERMOTRAUMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0033; 2019-A01163-54 (Other: ID-RCB)
Record Dates: First submitted 2019-05-15; First posted 2019-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Hypothermia; Trauma, Psychological
Keywords: body warmer; pre-hospital
MeSH Terms: conditions — Hypothermia; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ON (standard warming process + body warmer) (Experimental): Patients included during the ON periods will constitute the experimental group. Warming will be provided by the body warmer in addition to the standard warming procedure (survival blanket and heating in the emergency vehicle).
  Interventions: Device: Body warmer
- OFF / Control group (standard warming process ) (Sham Comparator): Patients included during the OFF periods will constitute the control group. Warming will be provided by the standard warming procedure : survival blanket and heating in the emergency vehicle.
  Interventions: Device: Standard warming procedure

INTERVENTIONS:
Device: Body warmer — The body warmer will be wrapped in a waterproof treatment field to avoid the risk of burns, 2 body warmer will be applied on the inguinal crease and 2 on the subclavicular fossa.
  Arms: ON (standard warming process + body warmer)
Device: Standard warming procedure — Warming only according to the standard procedure : survival blanket and heating in the emergency vehicle.
  Arms: OFF / Control group (standard warming process )

SUMMARY:
Study of adult patients with severe all-cause trauma having a body temperature less than 36°Celsius (C) that is managed by a Mobile Emergency Service team and oriented towards a Vital Emergency Room.

Currently two devices are used to warm patients during their care at the scene of an accident: a survival blanket and heating in the emergency vehicle. Despite these two devices many patients arrive in hypothermia (body temperature less than 36°C) in emergency departments. The objective of this study is to evaluate the effectiveness of a body warmer associated with standard warming devices on the correction of hypothermia compared to the standard procedure in severely traumatized patients with hypothermia .

It is a national multicentric study with 14 participating Mobile Emergency Service centers and hopefully will include 612 patients.

The study will be carried out according to a pattern of 28 successive periods of one week each during the winter period (October to April), for a total duration of 7 months. 14 action periods ON (warming standard procedure + body warmer) and 14 control periods OFF (warming standard procedure) will be run in random order for each center.

ELIGIBILITY:
Inclusion Criteria:

* Major patient with all-cause trauma Grade A or B
* Patient with a trans-tympanic body temperature of less than 36°Celsius (C) at primary management by terrestrial or heliport Mobile Emergency Service team.

Exclusion Criteria:

* Patient initially supported by a pre-hospital medical team who does not participate in the study,
* Patient with cardiopulmonary arrest at initial pre-hospital medical team management,
* Patient with bilateral otorrhagia (due to the non-feasibility of trans tympanic temperature),
* Patient with inguinal crease or subclavicular fossa injury,
* Patient with severe burn (Burnt Body Surface> 20%),
* Patient deprived of liberty including patients with an electronic bracelet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a temperature > 36°C when the patient arrived in the Vital Emergency | 4 hours
  Body temperature will be measured in trans-tympanic when the patient arrived in the Vital Emergency Room.

SECONDARY OUTCOMES:
Change in body temperature between initial treatment by the Mobile Emergency Service team and arrival at Vital Emergency Room. | 4 hours
  Body temperature will be measured in trans-tympanic every 15 minutes between initial treatment by the pre-hospital medical team and arrival at emergency room.
Proportion of patients with coagulopathy on arrival at the emergency room. | 4 hours
  Coagulopathy refers to disorders of blood coagulation whether they are pathological thrombosis or haemorrhagic syndromes. The coagulopathy criteria appear early and their measurements are systematically carried on admission to the emergency room.
Proportion of patients with acidosis on arrival at the emergency room. | 4 hours
  Acidosis is a disorder of the acid-base balance of the body corresponding to an increase in the concentration of acid in plasma and interstitial fluids. It can be metabolic or respiratory. In the case of a state of shock, lactic acid occurs in situations where the tissues of the body are poorly irrigated and lack oxygen.
Evaluation of mortality | 72 hours
  Proportion of deaths at one month (72h after admission to emergency room).
Evaluation of mortality (deaths before admission ) | 72 hours
  Proportion of deaths before admission to emergency room.
Evaluation of mortality (cardio respiratory arrest) | 72 hours
  Proportion of cardio respiratory arrest before admission to emergency room.
Loss of heat due to a drop of temperature | 4 hours
First degree burn | 4 hours
Patient feels cold | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Delphine HUGENSCHMITT, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- SAMU 69 - SMUR - Hôpital Edouard Herriot, Lyon, France